CLINICAL TRIAL: NCT04686604
Title: PRagmatic Trial Of Messaging to Providers About Treatment of Heart Failure in the Inpatient Setting
Acronym: PROMPT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2000029438; No NIH funding (Other: 10.11.23)
Record Dates: First submitted 2020-12-16; First posted 2020-12-29 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electron Health Record-based Provider Alert (Experimental): Providers will receive a best practice alert for each of their eligible patients upon opening of the order entry screen in the patient's medical record. The alert will inform the provider to the presence of HFrEF and of the patient's current left ventricular ejection fraction, most recent blood pressure and heart rate, most recent potassium and estimated glomerular filtration rate, and current evidence-based medications for HFrEF. It will also provide access to an order set with recommended evidence-based HFrEF therapies as well as a link to the best available guideline-recommended information regarding the treatment of heart failure.
  Interventions: Other: Best practice alert for the notification of patient HFrEF and recommended evidence-based medical therapies (NO drugs are being administered in this trial)
- Usual Care (No Intervention): Providers will not receive an alert and will proceed with usual care.

INTERVENTIONS:
Other: Best practice alert for the notification of patient HFrEF and recommended evidence-based medical therapies (NO drugs are being administered in this trial) — Providers will receive a best practice alert for each of their eligible patients upon opening of the order entry screen in the patient's medical record. The alert will inform the provider to the presence of HFrEF and of the patient's current left ventricular ejection fraction, most recent blood pressure and heart rate, most recent potassium and estimated glomerular filtration rate, and current evidence-based medications for HFrEF. It will also provide access to an order set with recommended evidence-based HFrEF therapies as well as a link to the best available guideline-recommended information regarding the treatment of heart failure.
  Arms: Electron Health Record-based Provider Alert

SUMMARY:
A randomized single-blind interventional trial to test the effectiveness of an electronic medical record-based best practice alert recommending evidence-based medical therapies versus usual care in inpatient adult patients presenting with heart failure with reduced ejection fraction.

DETAILED DESCRIPTION:
Heart failure (HF) is the major cause of healthcare expenditure, morbidity, and mortality in the United States. HF is the primary diagnosis for hospital discharge in ~1 million and a secondary diagnosis in ~2 million hospitalizations annually in the US. In fact, inpatient admissions account for more than half of HF healthcare expenditure. However, data from several registries over the last three decades has failed to see use of these evidence- based therapies at levels noted in clinical trials, despite aggressive guideline recommendations and promotion by thought leaders in the field. It remains unclear as to why many patients with HF reduced ejection fraction (HFrEF) are not on evidence-based therapies especially post hospital discharge and why the percentages are consistent across national registries over time. Whether the gap between clinical trial use and real-world practice is due to a lack of knowledge or providers making individualized decisions about their patients is unclear. A simple way to test this hypothesis is to examine whether electronic health record (EHR) based "best practice advisories" (BPAs) can increase use of evidence based therapies. If found to be effective, these low cost interventions can be rapidly applied across large healthcare systems.

The goal of this trial is to determine the effectiveness of a BPA alert system that informs providers about evidence-based medical therapy for the treatment of HFrEF versus usual care (no alert) in the inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years admitted to a hospital within the Yale New Haven Hospital system (either Yale New Haven Hospital, St. Raphael's Campus, Greenwich Hospital, or Bridgeport Hospital).
* Have HFrEF defined as:

  1. NT-pro-BNP >500 pg/ml within 24 hours of admission
  2. On IV loop diuretic within 24 hours of admission
  3. Left ventricular ejection fraction ≤40% (most recent)

Exclusion Criteria:

* Patients within 48 hours of admission
* Patients in the intensive care unit
* Patients on hospice service
* Patients receiving intravenous milrinone
* Patient on NPO (nothing by mouth) order
* Patients on all evidence based medical therapy for HFrEF (on all 4 classes of evidence based medical therapy: beta-blockers, ACEi/ARB/ARNI, MRA, SGLT2i)
* Opted out of medical record research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HFrEF with an increase in prescribed evidence-based HFrEF medical therapy | Assessed from the date of randomization to discharge date, assessed up to 12 months.
  Assessed as an increase in the number of prescribed targeted evidence-based medical therapies for HFrEF. Evidence-based medical therapies include: beta-blockers, ACEi/ARBs/ARNIs, MRAs, and SGLT2is.

SECONDARY OUTCOMES:
The percentage increase of beta blockers for HFrEF | Assessed from the date of randomization to discharge date, assessed up to 12 months.
  Increase in proportion of patients on beta blockers
The percentage increase of ACEi/ARB/ARNI for HFrEF | Assessed from the date of randomization to discharge date, assessed up to 12 months.
  Increase in proportion of patients on ACEi/ARB/ARNI
The percentage increase of MRAs for HFrEF | Assessed from the date of randomization to discharge date, assessed up to 12 months.
  Increase in proportion of patients on MRAs
The percentage increase of SGLT2i for HFrEF | Assessed from the date of randomization to discharge date, assessed up to 12 months.
  Increase in proportion of patients on SGLT2i
30-day hospital readmission rates | Assessed from the date of discharge to the date of hospital readmission, up to 30 days post-discharge
30-day emergency department visits | Assessed from the date of discharge to the date of ED/ER admission, up to 30 days post-discharge
6 months all-cause mortality | Assessed from the date of randomization to the date of death from any cause, up to 6 months post-randomization
Percentage of evidence-based medical therapy prescriptions for HFrEF filled by patients within 30 days of discharge | Assessed from the date of discharge and up to 30 days post-discharge.
  Percentage of patients who filled evidence-based medical therapies. Evidence-based medical therapies include: beta-blockers, ACEi/ARBs/ARNIs, MRAs, and SGLT2is.

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Ahmad, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data underlying results for publication will be made available upon publication of results.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication of results; indefinitely.

REFERENCES:
- [Derived] Ghazi L, O'Connor K, Yamamoto Y, Fuery M, Sen S, Samsky M, Riello RJ 3rd, Huang J, Olufade T, McDermott J, Inzucchi SE, Velazquez EJ, Wilson FP, Desai NR, Ahmad T. Pragmatic trial of messaging to providers about treatment of acute heart failure: The PROMPT-AHF trial. Am Heart J. 2023 Mar;257:111-119. doi: 10.1016/j.ahj.2022.12.002. Epub 2022 Dec 6. PMID 36493842
- See also: Trial Website — https://www.theprompttrials.org/